CLINICAL TRIAL: NCT06194409
Title: The Incidence, Clinical Characteristics and Outcome of Infective Endocarditis Among Intravenous Drug Abusers Versus Non-Drug Abusers.
Status: Recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Peter Alaa Adeab Eskarous, Resident at cardiology department, Faculty of medicine, Assiut University, Assiut University
Other Study IDs: Infective endocarditis
Record Dates: First submitted 2023-10-02; First posted 2024-01-08 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Infective Endocarditis
MeSH Terms: conditions — Endocarditis | interventions — Echocardiography; Urinalysis; Blood Culture

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- IE in IV drug abusers: Infective endocarditis in intravenous drug abusers
  Interventions: Diagnostic Test: Echocardiography, Urine analysis , blood culture
- IE in non- IV drug abusers: Infective endocarditis in non - intravenous drug abusers
  Interventions: Diagnostic Test: Echocardiography, Urine analysis , blood culture

INTERVENTIONS:
Diagnostic Test: Echocardiography, Urine analysis , blood culture — All patients will be investigated by ECG, Urine analysis, blood culture , Echocardiography

SUMMARY:
We aim to describe the incidence of IVDA among patients presented with IE, describe their clinical, psychiatric and microbiological characteristics in comparison to non - IVDA, as well as the rate and types of complications and outcome, and responsiveness to medical treatment or surgical intervention.

DETAILED DESCRIPTION:
Infective endocarditis (IE) is the infection of the endocardial surface of the heart mainly affecting the valves of the heart. It is still associated with very high morbidity and mortality all over the world despite various advances in diagnostic and treatment methods.

A few studies have shown that infective endocarditis represents less than 0.5% of adult cardiovascular admissions.While the overall incidence of IE has remained stable over the last several years, IE has increased in young people in parallel with injection drug use (IDU) behaviours and the growing opioid crisis.

According to recent guidelines , Intravenous (IV) drug use is considered a minor Duke criteria for the diagnosis of infective endocarditis.

Compared to the general population, intravenous drug abuse (IVDA) is associated with an up to 100-fold increased risk of IE through several mechanisms, including endothelial injury from injected particulate matter, direct injection of contaminated material, and drug-associated vasospasm leading to intimal damage and thrombus formation.

Also, IVDA is associated with HIV outbreaks, which is a well-known risk factor for IE. HIV-associated IE is associated with high rates of morbidity and mortality than non-HIV-associated IE.Because of its pathophysiology, IVDA-associated IE is more commonly right-sided. Beyond these known characteristics, however, literature on this topic is substantially limited, including the clinical and microbiological characteristics of these patients, rate and types of complications and outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adult Patients (>18 years) with definite or possible IE.

Exclusion Criteria:

* Patients with rejected diagnosis of infective endocarditis after workup, according to modified Duke's criteria.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients admitted to Assiut University Heart Hospital with definite or possible Infective endocarditis
Sampling Method: Non-Probability Sample
Enrollment: 46 (Estimated)
Dates: Start 2024-05-05 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
The incidence of IVDA among IE patients | Baseline
  Report the incidence of IVDA among IE patients, describe their clinical and microbiological characteristics comparison to the IE in non - IVDA.
The complications of IVDA among IE patients | Baseline
  Report the rates and types of complications

SECONDARY OUTCOMES:
The psychiatric characteristics of the addict group | Baseline
  This will be done by psychiatric questionnaires:
  -Addiction Severity Index questionnaire to measure severity of the addiction on the patient
The Withdrawal symptoms of the study group | Baseline
  This will be done by psychiatric questionnaires:
  -Withdrawal symptoms questionnaire that occur to the patient after stop of the addiction
The psychiatric characteristics of the study group | Baseline
  This will be done by psychiatric questionnaires:
  -Symptom Check List 90 to measure other comorbidities
The personality characteristics of the study group | Baseline
  This will be done by psychiatric questionnaires:
  -Eysenck Personality questionnaire to measure personality.

CONTACTS AND LOCATIONS:
Overall Officials: Yehia Kish, Study Director — Assiut University
Locations (1):
- Assiut University, Asyut, Egypt

REFERENCES:
- [Background] Math RS, Sharma G, Kothari SS, Kalaivani M, Saxena A, Kumar AS, Bahl VK. Prospective study of infective endocarditis from a developing country. Am Heart J. 2011 Oct;162(4):633-8. doi: 10.1016/j.ahj.2011.07.014. Epub 2011 Sep 14. PMID 21982654
- [Background] Noubiap JJ, Nkeck JR, Kwondom BS, Nyaga UF. Epidemiology of infective endocarditis in Africa: a systematic review and meta-analysis. Lancet Glob Health. 2022 Jan;10(1):e77-e86. doi: 10.1016/S2214-109X(21)00400-9. PMID 34919859
- [Background] Bor DH, Woolhandler S, Nardin R, Brusch J, Himmelstein DU. Infective endocarditis in the U.S., 1998-2009: a nationwide study. PLoS One. 2013;8(3):e60033. doi: 10.1371/journal.pone.0060033. Epub 2013 Mar 20. PMID 23527296
- [Background] Schranz AJ, Fleischauer A, Chu VH, Wu LT, Rosen DL. Trends in Drug Use-Associated Infective Endocarditis and Heart Valve Surgery, 2007 to 2017: A Study of Statewide Discharge Data. Ann Intern Med. 2019 Jan 1;170(1):31-40. doi: 10.7326/M18-2124. Epub 2018 Dec 4. PMID 30508432
- [Background] Delgado V, Ajmone Marsan N, de Waha S, Bonaros N, Brida M, Burri H, Caselli S, Doenst T, Ederhy S, Erba PA, Foldager D, Fosbol EL, Kovac J, Mestres CA, Miller OI, Miro JM, Pazdernik M, Pizzi MN, Quintana E, Rasmussen TB, Ristic AD, Rodes-Cabau J, Sionis A, Zuhlke LJ, Borger MA; ESC Scientific Document Group. 2023 ESC Guidelines for the management of endocarditis. Eur Heart J. 2023 Oct 14;44(39):3948-4042. doi: 10.1093/eurheartj/ehad193. No abstract available. PMID 37622656
- [Background] Scheggi V, Del Pace S, Ceschia N, Vanni F, Merilli I, Sottili E, Salcuni L, Zoppetti N, Alterini B, Cerillo A, Marchionni N, Stefano PL. Infective endocarditis in intravenous drug abusers: clinical challenges emerging from a single-centre experience. BMC Infect Dis. 2021 Sep 27;21(1):1010. doi: 10.1186/s12879-021-06697-1. PMID 34579674
- [Background] Goyal A, Mohan B, Kumar P, Gupta D, Tandon R, Singla S, Singh G, Singh B, Chhabra ST, Aslam N, Wander GS. Clinical characteristics and outcome of infective endocarditis among intravenous drug abusers in India. Indian Heart J. 2020 Nov-Dec;72(6):547-551. doi: 10.1016/j.ihj.2020.09.014. Epub 2020 Sep 18. PMID 33357643
- [Background] McLellan AT, Luborsky L, Woody GE, O'Brien CP. An improved diagnostic evaluation instrument for substance abuse patients. The Addiction Severity Index. J Nerv Ment Dis. 1980 Jan;168(1):26-33. doi: 10.1097/00005053-198001000-00006. PMID 7351540
- [Background] Derogatis, L.R. and Savitz, K.L. (2000) The SCL-90-R and the Brief Symptom Inventory (BSI) in Primary Care. In:: Maruish, M.E., Ed., Handbook of Psychological Assessment in Primary Care Settings, Vol. 236, Lawrence Erlbaum Associates, Mahwah, 297-334
- [Background] Hans Jürgen Eysenck & Sybil B. G. Eysenck (1975). Manual of the Eysenck Personality Questionnaire, London: Hodder and Stoughton
- [Background] Macingwane J., Ngwenya B.N. Identification of active compounds of Albizia lebbeck against HIV-1 reverse transcriptase: a computational study. J. Biomol. Struct. Dyn. 2021;39(14):5300-5311. [Google Scholar]